CLINICAL TRIAL: NCT04721873
Title: Pharmacologic Weight Loss as Adjunct Therapy for Ulcerative Colitis in Obese Patients: A Phase 2A, Randomized, Placebo-Controlled Trial
Brief Title: Pharmacologic Weight Loss as Adjunct Therapy for Ulcerative Colitis in Obese Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Siddharth Singh, Assistant Professor of Medicine, Division of Gastroenterology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 190419; 623346 (Other Grant/Funding Number: Litwin Pioneers in IBD, Crohn's and Colitis Foundation)
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Colitis, Ulcerative; Obesity
MeSH Terms: conditions — Colitis, Ulcerative; Obesity | interventions — Qsymia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: Phentermine-Topiramate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phentermine-Topiramate — Patients will be randomized to either once-daily, oral phentermine-topiramate 15-92mg or placebo, in a 1:1 fashion, for 22 weeks, with clinic visits with an obesity medicine specialist, for intensive counseling for diet and lifestyle intervention. All patients will be dose-titrated within the first 4 weeks, starting at phentermine-topiramate 3.75-23mg, or placebo. Dose titration will be performed as follows 3.75-23mg x 1 week --> 7.5-46mg x 1 week --> 11.25-69mg x 1 week --> 15-92mg. Patients who experience side effects would undergo slower titration, and dose would be down-titrated and capped at highest tolerated dose.
  Arms: Intervention
Drug: Placebo — Matching placebo, titrated as active intervention
  Arms: Placebo

SUMMARY:
Approximately 20-40% of patients with ulcerative colitis (UC) are obese. The investigators have demonstrated that obesity adversely impacts disease course in patients with UC, leading to higher risk of persistently active disease, surgery, hospitalization, and treatment failure, particularly in biologic-treated patients. Intentional weight loss is effective in improving disease outcomes in patients with inflammatory arthritis, but there is limited data on its impact in UC. While dietary interventions for weight loss have limited efficacy and endoscopic bariatric interventions may be too invasive in patients with UC with active gastrointestinal symptoms, pharmacological weight loss with a highly effective oral agent may be a novel strategy to induce weight loss and augment the efficacy of biologic therapy in UC.

Hence, the investigators are conducting a pilot, phase 2A, 22-week, randomized, placebo-controlled clinical trial of phentermine-topiramate in obese patients with active UC starting on a new biologic agent (infliximab, adalimumab, golimumab, vedolizumab).

The overall objective is to (1) evaluate the efficacy, safety and tolerability of phentermine-topiramate, and (2) to assess the impact of pharmacological weight loss on clinical outcomes, inflammatory burden and biologic trough concentration in patients with UC. The central hypothesis is that phentermine-topiramate will be safe, effective, and well tolerated in patients with UC, and weight loss would achieve higher rates of clinical and biochemical remission, and higher biologic trough concentration.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-80y
* BMI ≥30kg/m^2
* established diagnosis of UC based on clinical and endoscopy evidence corroborated by histopathology report
* active UC (Mayo Clinic score [MCS], 6-12; or active disease based on rectal bleeding score [RBS]=2 or 3 and stool frequency score=2 or 3) or dependent on corticosteroids (unable to taper below 10mg prednisone equivalent, or flaring within 2 months of stopping prednisone)
* starting a new biologic agent (TNFα antagonists, vedolizumab, ustekinumab) or flaring despite stable maintenance dose of biologic agent
* stable weight (<5kg weight change) for preceding 4 weeks prior to screening and randomization
* able to speak or understand English and provide written informed consent.

Exclusion Criteria:

* pregnant or lactating women
* prisoners
* current or history of toxic megacolon, abdominal abscess, symptomatic intestinal or colonic stricture, history of colectomy or diverting stoma, short bowel syndrome, active tuberculosis or other bacterial infections, cancer
* any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise patient safety
* clinically meaningful laboratory abnormalities, including significant anemia (Hb<8g/dl), leukopenia (<3x10^9/L), thrombocytopenia (<100K) or thrombocytosis (>600K), ALT/AST >3x upper limit of normal, creatinine >2x upper limit of normal
* blood pressure >140/95mmHg (ok to include if BP controlled on anti-hypertensives), fasting blood glucose >240mg/dl or HbA1c >9%, fasting triglycerides >400mg/dl at randomization, type 1 diabetes, coronary artery disease, stroke, or other symptomatic peripheral arterial disease
* history of nephrolithiasis (H/O kidney stone >1 time, and kidney stone within 1y prior to start of study), hyperthyroidism, seizure disorder
* recurrent major depression, presence or history of suicidal behavior or ideation with intent to act, current substantial depressive symptoms (patient health questionnaire-9, ≥10), use of antidepressant medication that has not been stable for the prior 3 months (bupropion-treated patients will be excluded)
* history of (or treatment for) glaucoma or increased intraocular pressure
* prior bariatric surgery; >5 kg weight fluctuation in preceding 4 weeks, use of very-low-calorie diet, or participation in a formal weight loss program in the 3 months prior to the study
* smoking cessation within previous 3 months or plans to quit during the study period
* history of eating disorder or drug/alcohol abuse within the preceding 1 year concomitant use of other sympathomimetic medications, for example for ADHD
* known allergy to study medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight loss - 5% | 22 weeks
  Proportion of patients with ≥5% weight loss over baseline

SECONDARY OUTCOMES:
Weight loss - 10% | 22 weeks
  Proportion of patients with ≥10% weight loss over baseline
Absolute weight loss | 22 weeks
  Absolute weight loss from baseline
Discontinuation | 22 weeks
  Discontinuation of therapy due to treatment-related adverse events
Corticosteroid-free clinical remission | 22 weeks
  PRO2 remission, with no prednisone use within 1 week of assessment
Biochemical remission | 22 weeks
  Fecal calprotectin (FC) ≤50μg/g

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided